CLINICAL TRIAL: NCT03525106
Title: Feasibility of a Positive Psychology Intervention for Hematopoietic Cell Transplant Survivors to Improve Quality of Life
Brief Title: Positive Psychology Intervention to Improve Quality of Life in Stem Cell Transplant Survivors and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9969; NCI-2018-00541 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9969 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2018-04-17; First posted 2018-05-15 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Hematopoietic Cell Transplantation Recipient

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants: Positive Psychology Intervention (Experimental): Participants receive a positive psychology exercise manual, complete positive psychology exercises every week, and participate in phone sessions over 30 minutes every week for 8 weeks.
  Interventions: Behavioral: Booklet; Behavioral: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Survey Administration; Behavioral: Telephone-Based Intervention
- Caregivers: Positive Psychology Intervention (Experimental): Caregivers receive a positive psychology exercise manual, complete positive psychology exercises every week, and participate in phone sessions over 30 minutes every week for 8 weeks.
  Interventions: Behavioral: Booklet; Behavioral: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Survey Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Behavioral: Booklet — Receive positive psychology manual
  Other Names: Pamphlet
Behavioral: Exercise Intervention — Complete positive psychology exercises
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Participate in phone sessions

SUMMARY:
This trial studies a positive psychology intervention designed to improve quality of life in stem cell transplant survivors and their caregivers. Positive psychology (PP) uses systematic exercises (e.g., gratitude letters, acts of kindness) to potentially boost levels of optimism, resilience, and life enjoyment. PP interventions are often enjoyable, easy to understand, and can be delivered via telephone. PP intervention may improve the quality of life of participants who have undergone a stem cell transplant or their caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Pilot a positive psychology intervention delivered to hematopoietic cell transplantation (HCT) survivors and interested caregivers over an 8 week period.

II. Determine the proportion of patients who enroll and the immediate benefit to participants, as measured by pre- and post-exercise measures of happiness and optimism.

III. Pilot outcome data collection mechanisms in preparation for a randomized clinical trial.

OUTLINE:

Participants and caregivers receive a positive psychology exercise manual, complete positive psychology exercises every week, and participate in phone sessions over 30 minutes every week for 8 weeks.

After completion of study, participants are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* English as primary language
* At least 1 year after HCT

Exclusion Criteria:

* Major psychiatric diagnosis that impairs cognitive functioning or is not controlled at the time of the approach.
* Medical conditions precluding participation in the intervention or likely to lead to death within 6 months, as determined by the principal investigator (PI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Study enrollment rates | Up to 8 weeks
  The analysis of the study will mainly be descriptive. The proportion of participants who consent to enroll in the study will be computed based on the number approached through each method. Reasons for non-participation will be summarized. A larger randomized trial will be considered feasible if the enrollment rate for patients approached in person or over the phone is > 50% (excluding the active opt-out rate) and the overall completeness of follow-up data collection is > 70%, excluding patients who have died or are hospitalized/ill at the assessment point.
  Since the number of caregivers who will participate is unknown, caregiver analyses will also be descriptive only.
Positive psychology intervention completion rates | Up to 8 weeks
Completeness of follow-up data collection | Up to 8 weeks
  Completeness is defined by the proportion of instrument scores that can be calculated per given time point. The completeness of follow-up data collection will be calculated and reported as a proportion of successfully completed scales versus scales attempted to be collected or completed by patients.
Changes in happiness after each exercise | Baseline up to 8 weeks
  Change in happiness for each exercise will be analyzed by change scores. A change of 2 points on a 0-10 scale, with 10 being happiest, is considered clinically meaningful.
Changes in optimism after each exercise | Baseline up to 8 weeks
  Change in optimism for each exercise will be analyzed by change scores. A change of 2 points on a 0-10 scale, with 10 being most optimistic, is considered clinically meaningful.
Changes in mental health | Baseline up to 6 months after intervention ends
  This will be assessed with the patient-reported outcomes measurement information system, PROMIS-10 (Global-Mental). Higher scores are better. T scores will be used to standardize scores so that 50 represents the US general population and 10 is the standard deviation.
Changes in physical health | Baseline up to 6 months after intervention ends
  This will be assessed with the patient-reported outcomes measurement information system, PROMIS-10 (Global-Physical). Higher scores are better. T scores will be used to standardize scores so that 50 represents the US general population and 10 is the standard deviation.
Changes in fatigue | Baseline up to 6 months after intervention ends
  This will be assessed with the patient-reported outcomes measurement information system, PROMIS-Fatigue. Lower scores are better. T scores will be used to standardize scores so that 50 represents the US general population and 10 is the standard deviation.
Changes in pain | Baseline up to 6 months after intervention ends
  This will be assessed with the patient-reported outcomes measurement information system, PROMIS-Pain interference. Lower scores are better. T scores will be used to standardize scores so that 50 represents the US general population and 10 is the standard deviation.
Changes in resilience | Baseline up to 6 months after intervention ends
  This will be assessed with the Connor Davidson resilience scale. Total scores range from 0-40 with higher scores reflecting great resilience.
Changes in anxiety and depression | Baseline up to 6 months after intervention ends
  The Hospital Anxiety and Depression Scale will be used to capture depression and anxiety. Scores on the Anxiety and Depression subscales range from 0-21 with higher scores indicating more distress. Subscales will be reported separately.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States